CLINICAL TRIAL: NCT02543645
Title: A Phase l/ll, Open Label, Dose-escalation Study of Varlilumab (CDX-1127) in Combination With Atezolizumab (MPDL3280A, Anti-PD-L1) in Patients With Advanced Cancer
Brief Title: A Study of Varlilumab and Atezolizumab in Patients With Advanced Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Portfolio re-prioritization
Sponsor: Celldex Therapeutics (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDX1127-06
Record Dates: First submitted 2015-08-28; First posted 2015-09-07 (Estimated); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Carcinoma, Renal Cell; Kidney Diseases; Kidney Neoplasms; Urogenital Neoplasms; Urologic Diseases; Urologic Neoplasms; Neoplasms by Histologic Type; Neoplasms; Clear-cell Metastatic Renal Cell Carcinoma; Melanoma; Triple Negative Breast Cancer; Bladder Cancer; Head and Neck Cancer; Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Diseases; Kidney Neoplasms; Urogenital Neoplasms; Urologic Diseases; Urologic Neoplasms; Neoplasms by Histologic Type; Neoplasms; Clear-cell metastatic renal cell carcinoma; Melanoma; Triple Negative Breast Neoplasms; Urinary Bladder Neoplasms; Head and Neck Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Varlilumab and Atezolizumab (Experimental)
  Interventions: Drug: Combination of Varlilumab and Atezolizumab

INTERVENTIONS:
Drug: Combination of Varlilumab and Atezolizumab — Treatment cycles are 12 weeks each with varlilumab and atezolizumab administered every 3 weeks. During the treatment phase of the study, eligible patients will receive varlilumab for up to 3 cycles (with a 4th cycle possible following discussion with the Medical Monitor). There is no limit on the number of cycles of atezolizumab. Patients may be discontinued from receiving study treatment (atezolizumab or varlilumab) based on the results of disease assessments or if experiencing side effects that make study therapy intolerable.
  Phase l Dose: The planned dose of varlilumab will be dependent on the cohort assigned at enrollment. Varlilumab doses are 0.3 mg/kg, 1 mg/kg, or 3 mg/kg. The dose of atezolizumab is 1200 mg.

SUMMARY:
This is a study to determine the clinical benefit (how well the drug works), safety and tolerability of combining varlilumab and atezolizumab. Phase l of the study will enroll patients with a number of tumor types; Phase ll will enroll only patients with renal cell carcinoma (RCC).*

*Note: This Study was terminated prior to initiation of Phase II

DETAILED DESCRIPTION:
Varlilumab is a fully human monoclonal antibody that binds to a molecule called CD27 found on certain immune cells and may act to promote anti-tumor effects.

Atezolizumab is an engineered anti-PD-L1 antibody.

This study will evaluate the safety, tolerability and efficacy of the anti-CD27 antibody varlilumab in combination with atezolizumab.

Eligible patients that enroll in the dose escalation portion of the study will be assigned to one of three dose levels of varlilumab in combination with 1200 mg of atezolizumab. The first phase of the study will enroll up to 18 patients and test the safety profile of the combination of varlilumab and atezolizumab in patients with various tumor types and determine which dose of varlilumab will be studied in Phase ll* of the study which will enroll only patients with RCC.

*Note: This Study was terminated prior to initiation of Phase II.

All patients enrolled in the study will be closely monitored to determine if there is a response to the treatment as well as for any side effects that may occur.

ELIGIBILITY:
Inclusion Criteria:

1. Unresectable stage lll or IV, histologically confirmed diagnosis of one of the following solid tumors:

   * Phase l: Melanoma, RCC, triple negative breast cancer, bladder cancer, head and neck cancer or non-small cell lung cancer.
2. Documented progressive disease based on radiographic, clinical or pathologic assessment during or subsequent to last therapy.
3. Progressed or intolerant to at least 1 approved prior anticancer regimen.
4. Measurable (target) disease.
5. Life expectancy ≥ 12 weeks.
6. If of childbearing potential (male or female), agrees to practice an effective form of contraception during study treatment and for at least 90 days following last treatment dose.
7. Must have available tumor tissue and consent to biopsy while on study.
8. Patients with asymptomatic treated CNS metastasis may be enrolled after discussion with the Medical Monitor.
9. ECOG of 0 or 1.

Exclusion Criteria:

1. Prior therapy with varlilumab or with an anti-CD27 antibody.
2. Previous treatment with anti-PD-1, anti-PD-L1 or anti-PD-L2 therapy.
3. Use of any experimental immunotherapy.
4. Receipt of anti-CTLA-4 targeted therapies or other checkpoint or co-stimulatory therapy within 3 months prior to start of study treatment.
5. Chemotherapy within 21 days or at least 5 half-lives (whichever is shorter) prior to the planned state of study treatment.
6. Systemic radiation therapy within 4 weeks, prior focal radiotherapy within 2 weeks, or radiopharmaceuticals (strontium, samarium) within 8 weeks prior to the first dose of study treatment.
7. Use of immunosuppressive medications within 4 weeks or systemic corticosteroids within 2 weeks prior to first dose of study treatment.
8. Other prior malignancy, except for adequately treated basal or squamous cell skin cancer or in situ cancers; or any other cancer from which the patient has been disease-free for at least 3 years.
9. Active, untreated CNS metastases.
10. Active autoimmune disease or a documented history of autoimmune disease.
11. Active diverticulitis.
12. Significant cardiovascular disease including CHF, leptomeningeal disease, poorly controlled hypertension, or an MI within 6 months prior to dosing.
13. Known alcohol or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-10; Primary Completion 2017-04 (Actual); Study Completion 2017-05-22 (Actual)

PRIMARY OUTCOMES:
Phase l: Safety and tolerability of varlilumab in combination with atezolizumab as measured by incidence of drug related adverse events (AEs), serious drug related AEs, dose-limiting toxicities and laboratory test abnormalities. | Safety follow-up is 70 days from last study drug dose.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of California - San Francisco, San Francisco, California
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina